CLINICAL TRIAL: NCT03902496
Title: Optical Treatment of Migraines Clinical Study
Brief Title: Optical Treatment of Migraines Using the Avulux™ Optical Filter in the Form of Spectacle Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avulux, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20190592
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: A total of 50 subjects will be randomized into one of two treatment groups in a one-to-one ratio. After three weeks, and following a one-week washout period, subjects will be given spectacles from the other treatment group
Who Masked: Participant, Care Provider, Investigator
Masking Description: The active and sham lenses will have tints calibrated such that the optical density, that is the overall "darkness" of all study lenses, will be the same. All study lenses will appear to have the same overall light-blocking effect to study subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Avulux Spectacles (Experimental): Subjects will be instructed to use the spectacles for three weeks. They will be instructed to put the spectacles on at the first signs or symptoms of their migraine attacks. This could be their usual aura, or the first signs of their headache commencing, and to keep the spectacles on until their headache has resolved.
  Interventions: Other: HIT-6 Questionnaire; Device: Avulux Spectacles
- Sham Spectacles (Sham Comparator): Subjects will be instructed to use the spectacles for three weeks. They will be instructed to put the spectacles on at the first signs or symptoms of their migraine attacks. This could be their usual aura, or the first signs of their headache commencing, and to keep the spectacles on until their headache has resolved.
  Interventions: Other: HIT-6 Questionnaire; Device: Sham Spectacles

INTERVENTIONS:
Other: HIT-6 Questionnaire — Headache Impact Test
Device: Avulux Spectacles — Avulux™ Optical Filter in the Form of Spectacle Lenses
  Arms: Avulux Spectacles
Device: Sham Spectacles — Sham
  Arms: Sham Spectacles

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the Avulux device in reducing the impact of migraine headaches as measured by improvement in Headache Impact Test (HIT-6TM) scores at three weeks when compared to a control/sham device.

DETAILED DESCRIPTION:
Avulux™ is intended to decrease the impact of headache and migraine on normal daily life and the ability to function, and reduce the frequency and severity of headache, in adult patients diagnosed with episodic migraine headache or chronic migraine.

Avulux™ consists of a pair of optical filters in the form of spectacle lenses, provided in standard spectacle frames or as clip-on units, coated with a thin film that effectively blocks light at specified wavelength ranges while minimizing distortion of the visible spectrum. The optical filters block a portion of the optical spectrum that is suspected to stimulate photophobic responses that trigger some, and exacerbate most, migraines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years or older
2. Patient is willing and able to provide written informed consent
3. Patient is willing and able to complete all scheduled study visits
4. Diagnosis of migraine, based on the following primary headache characteristics:

   1. At least 5 attacks fulfilling criteria b-d:
   2. Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
   3. Headache has at least two of the following characteristics:

      * unilateral location
      * pulsating quality
      * moderate or severe pain intensity
      * aggravation by or causing avoidance of routine physical activity (eg, walking or climbing stairs)
   4. During headache at least one of the following:

      * nausea and/or vomiting
      * photophobia and phonophobia
   5. Not attributed to another disorder

Exclusion Criteria:

1. Patients with other light sensitive conditions, such as iritis.
2. Patients who have less than 4 headache days per month
3. Patients who have chronic daily headaches.
4. Patients who have had any change in their migraine treatment within the 4 weeks prior to the trial onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test (HIT-6) total score | Three-week
  The primary objective of this study is to evaluate the efficacy of the Avulux device in reducing the impact of migraine headaches as measured by improvement in Headache Impact Test (HIT-6) scores at three weeks when compared to a control/sham device. HIT-6 scores range from 36 to 78. Higher scores indicate a greater impact of headaches on the respondent's life, i.e., 36 = no impact, 78 = maximum impact.

SECONDARY OUTCOMES:
Number and Severity of Headache Days | Three-week
  To measure effects on the number and severity of headaches, we will use the subjects' daily diaries to count the number of days with headache that either a) made activity difficult, b) caused activity changes, or c) caused patient to go to bed. We will then compare the proportion of days with headaches that met one of these criteria for the 4-week baseline period and the 3-week intervention.

OTHER OUTCOMES:
Proportion of subjects who were able to move out of the "very severe impact" category of the HIT-6 during the 3-week intervention | Three-week
  Compare initial vs. final HIT-6 scores for each treatment period
Proportion of patients who experienced at least a 5-point improvement in their HIT-6 score during the 3-week intervention | Three-week
  Compare initial vs. final HIT-6 scores for each treatment period
Proportion of days with headaches which lead to use of medications to control the headache over the 3-week intervention | Three-week
  Compare diaries for treatment vs. control periods to determine proportion of headaches resolved by device vs. device plus medication
Proportion of days with light sensitivity over the 3-week intervention | Three-week
  Compare diaries for treatment vs. control periods to determine differences in days with light sensitivity.
Average Number of Hours Slept over the 3-week intervention | Three-week
  Compare diaries for treatment vs. control periods to determine whether a significant difference exists in number of hours slept between treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Remington-Davis Clinical Research, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT03902496/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT03902496/ICF_001.pdf